CLINICAL TRIAL: NCT03035045
Title: Oral Paracetamol Premedication Effect on Maternal Pain in Amniocentesis: A Randomized Double Blind Placebo-controlled Trial
Brief Title: Oral Paracetamol Premedication Effect on Maternal Pain in Amniocentesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RJPARA
Record Dates: First submitted 2016-11-16; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-11

CONDITIONS: Amniocentesis
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Comparator1: Paracetamol 650 mg (325 mg/tablet) oral (Experimental): Drug: Paracetamol Comparison pain score between paracetamol and placebo
  Interventions: Drug: Paracetamol
- Comparator 2: Placebo oral (Placebo Comparator): Drug: placebo Comparison pain score between paracetamol and placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Paracetamol
  Arms: Comparator1: Paracetamol 650 mg (325 mg/tablet) oral
Drug: Placebo Oral Tablet
  Arms: Comparator 2: Placebo oral

SUMMARY:
This randomized controlled trial, compares perioperative and postoperative pain score by using visual analog scale in pregnant women undergoing amniocentesis. The experimental group will be given oral paracetamol premedication whereas the controlled group will be given oral placebo premedication.

DETAILED DESCRIPTION:
Perioperative and postoperative amniocentesis are often painful which cause concerns to those who has to undergo amniocentesis. Anxiety is one of the factor that may prolong operative time, resulting in an increase risk of complication from the procedure. Furthermore, pregnant women, in order to relief the pain, might require others drugs, which has both maternal and fetal side effect. So In conclusion, this study aims to compare efficacy of oral paracetamol premedication and oral placebo premedication by using visual analog scale to evaluate pain.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnant women undergo amniocentesis for the first time at Rajavithi Hospital in 2016-2017

Exclusion Criteria:

* Pregnant women with psychiatric disorder
* Contraindicated to paracetamol
* Pregnant women undergoing amniocentesis due to fetal anomaly
* Take oral paracetamol or other analgesics within 24-48 hrs before operation
* Deny to participate the research

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Different in pain score on visual analog scale in amniocentesis between controlled group (placebo) and experimental group (paracetamol). | 1 yrs

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Bangkok, Thailand